CLINICAL TRIAL: NCT06403761
Title: Effect of CagriSema, Semaglutide and Cagrilintide on Insulin Sensitivity and Pancreatic Endocrine Function in Adults With Type 2 Diabetes
Brief Title: Investigating How CagriSema, Semaglutide and Cagrilintide Regulate Insulin Effects in the Body of People With Type 2 Diabetes
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9388-7782; U1111-1300-1930 (Other: World Health Organization (WHO)); 2023-509483-20 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide; cagrilintide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CagriSema (Experimental): Participants will receive once-weekly subcutaneous (s.c) injections of CagriSema (cagrilintide and semaglutide) at escalating doses every 4 weeks in a 16-week dose escalation period until target dose of CagriSema is achieved and maintained for 12 weeks.
  Interventions: Drug: Semaglutide; Drug: Cagrilintide; Drug: Placebo semaglutide; Drug: Placebo cagrilintide
- Semaglutide (Experimental): Participants will receive once-weekly s.c injections of semaglutide at escalating doses every 4 weeks in a 16-week dose escalation period until target dose of CagriSema is achieved and maintained for 12 weeks.
  Interventions: Drug: Semaglutide; Drug: Placebo semaglutide
- Cagrilintide (Experimental): Participants will receive once-weekly s.c injections of cagrilintide at escalating doses every 4 weeks in a 16-week dose escalation period until target dose of CagriSema is achieved and maintained for 12 weeks.
  Interventions: Drug: Cagrilintide; Drug: Placebo cagrilintide
- Placebo (Placebo Comparator): Participants will receive once-weekly s.c injection of placebo matched to semaglutide and cagrilintide for 28 weeks.
  Interventions: Drug: Placebo semaglutide; Drug: Placebo cagrilintide

INTERVENTIONS:
Drug: Semaglutide — Participants will receive once-weekly semaglutide subcutaneously.
  Arms: CagriSema; Semaglutide
Drug: Cagrilintide — Participants will receive once-weekly cagrilintide subcutaneously.
  Arms: CagriSema; Cagrilintide
Drug: Placebo semaglutide — Participants will receive once-weekly placebo matched to semaglutide subcutaneously.
  Arms: CagriSema; Placebo; Semaglutide
Drug: Placebo cagrilintide — Participants will receive once-weekly placebo matched to cagrilintide subcutaneously.
  Arms: CagriSema; Cagrilintide; Placebo

SUMMARY:
This study will look at how CagriSema, semaglutide and cagrilintide regulate insulin effects in the body of people with type 2 diabetes (T2D). CagriSema is a new investigational medicine that combines two medicines called cagrilintide and semaglutide. Doctors may not yet prescribe CagriSema. Participants will either get CagriSema, semaglutide, cagrilintide, or a ''dummy'' medicine. Which treatment the participants will get is decided by chance. Participants will get the study medicine together with the current daily diabetes medicine metformin. Participants should not take other medicines for diabetes during the study. The study will last for about 42 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Aged 18-75 years (both inclusive) at the time of signing informed consent.
* Diagnosed with type 2 diabetes greater than or equal to (>=) 180 days before screening.
* Stable daily dose(s) of metformin at effective or maximum tolerated dose, as judged by the investigator for 90 or more days before screening with or without one additional oral antidiabetic drug (OAD), except for the use of glucagon-like peptide-1 (GLP-1) receptor agonists, or sodium-glucose co-transporter-2 (SGLT-2) inhibitors in case of a high risk of cardiovascular disease (as judged by the investigator), or established cardiovascular disease, or chronic kidney disease (Glomerular Filtration Rate (eGFR) less than (<) 60 milliliter per minute per 1.73 square meter [ml/min/1.73 m^2]).
* Glycated hemoglobin (HbA1c) at screening of 6.5-9.5 percent (48-80 millimoles per mole [mmol/mol]) (both inclusive) if on metformin only, or 6.0- 9.0 percent (42-75 mmol/mol) (both inclusive) if on metformin in combination with one other OAD. A minimum of 65% of randomised participants must have HbA1c >= 7.0 % at screening.
* Body Mass index (BMI) between 25.0 and 45.0 kilogram per square meter (kg/m^2) (both inclusive) at screening.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using highly effective contraceptive method.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* Renal impairment with estimated Glomerular Filtration Rate (eGFR) < 45 ml/min/1.73 m^2 at screening.
* Treatment with any medication for the indication of T2D or weight management other than stated in the inclusion criteria within 90 days before screening. However, short term insulin treatment for a maximum of 14 consecutive days and prior insulin treatment for gestational diabetes are allowed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-02-13 (Estimated)

PRIMARY OUTCOMES:
To compare the effect of CagriSema versus placebo: Change in M-value in hyperinsulinaemic euglycaemic clamp (HEC) | Baseline to week 28
  M-value from the HEC is calculated from glucose infusion rate (GIR) over the last 30 minutes of the clamp, corresponding to steady state. M-value is defined as: (GIR150-180 min normalised by body weight [milligram per minute per kilogram {mg/min/kg}]). Measured in mg/min/kg.

SECONDARY OUTCOMES:
To compare the effect of CagriSema versus semaglutide, Semaglutide versus placebo and Cagrilintide versus placebo: Change in M-value in HEC | Baseline to week 28
  M-value from the HEC is calculated from GIR over the last 30 minutes of the clamp, corresponding to steady state. M-value is defined as: (GIR150-180 min normalised by body weight [mg/min/kg]). Measured in mg/min/kg.
To compare the effect of CagriSema versus placebo, CagriSema versus semaglutide, Semaglutide versus placebo and Cagrilintide versus placebo: Change in M-value in HEC, normalised by lean body mass | Baseline to week 28
  M-value from the HEC is calculated from GIR over the last 30 minutes of the clamp, corresponding to steady state. M-value is defined as: (GIR150-180 min normalised by body weight [mg/min/kg]). Measured in mg/min/kg.
Change in first-phase incremental insulin secretion rate (ISR0-8min) in hyperglycaemic clamp (HGC) | Baseline to week 28
  Measured in picomoles per minute per square meter (pmol/min/m^2).
Change in second-phase insulin secretion rate (ISR20-120min) in HGC | Baseline to week 28
  Measured in pmol/min/m^2.
Change in total insulin secretion rate (ISR0-120min) in HGC | Baseline to week 28
  Measured in pmol/min/m^2.
Change in insulin secretion rate at fixed glucose concentration (ISRg) in HGC | Baseline to week 28
  Measured in pmol/min/m^2.
Change in total insulin response (total AUC0-120 min) in HGC | Baseline to week 28
  Measured in minute * picomoles per liter (min*pmol/L).
Change in insulin response to arginine (incremental insulin AUCarginine,0-10min) in HGC | Baseline to week 28
  Measured in min*pmol/L.
Change in C-peptide response to arginine (incremental insulin AUCarginine,0-10min) in HGC | Baseline to week 28
  Measured in min*nmol/L.
Change in clamp disposition index (cDI) calculated from HEC and HGC | Baseline to week 28
  cDI is defined as the product of the M-value derived from the hyperinsulinemic euglycemic clamp over the last 30 minutes and total insulin secretion (ISR AUC0-120min) derived from the insulin secretion rate based on C-peptide using the using the deconvolution technique divided by the total glucose AUC0-120min from the hyperglycemic clamp portion of the study. Measured in picomoles * liter per square meter per square minute per kilogram (pmol*L/m^2/min^2/kg).
Change in cDI calculated from HEC and HGC,based on lean body mass | Baseline to week 28
  cDI is defined as the product of the M-value derived from the hyperinsulinemic euglycemic clamp over the last 30 minutes and total insulin secretion (ISR AUC0-120min) derived from the insulin secretion rate based on C-peptide using the using the deconvolution technique divided by the total glucose AUC0-120min from the hyperglycemic clamp portion of the study. Measured in pmol*L/m^2/min^2/kg.
Change in β-cell glucose sensitivity (insulin secretion) from HGC | Baseline to week 28
  Measured in picomoles per minute per square meter per millimoles per liter (pmol/min/m^2/[mmol/L]).
Change in β-cell glucose sensitivity from mixed meal tolerance test (MMTT) (slope of dose-response for insulin secretion vs. plasma glucose) | Baseline to week 28
  Measured in pmol/min/m^2/(mmol/L).
Change in glucose concentration during MMTT (total and incremental AUC0-300min) | Baseline to week 28
  Measured in minute * millimoles per liter (min*mmol/L).
Change in insulin concentration during MMTT (total and incremental AUC0-300min) | Baseline to week 28
  Measured in minute * picomoles per liter (min*pmol/L).
Change in C-peptide concentration during MMTT (total and incremental AUC0-300min) | Baseline to week 28
  Measured in minute * nanomole per liter (min*nmol/L).
Change in glucagon concentration during MMTT (total and incremental AUC0-300min) | Baseline to week 28
  Measured in min*pmol/L.
Change in fasting glucose concentration (MMTT pre-meal concentrations) | Baseline to week 28
  Measured in millimole per liter (mmol/L).
Change in fasting insulin concentration (MMTT pre-meal concentrations) | Baseline to week 28
  Measured in picomole per milliliter (pmol/mL)
Change in fasting C-peptide concentration (MMTT pre-meal concentrations) | Baseline to week 28
  Measured in nanomoles per liter (nmol/L).
Change in fasting glucagon concentration (MMTT pre-meal concentrations) | Baseline to week 28
  Measured in picomoles per liter (pmol/L).
Change in fasting proinsulin concentration (MMTT pre-meal concentrations) | Baseline to week 28
  Measured in pmol/L.
Change in HbA1c | Baseline to week 28
  Measured as percentage points (%-points).
Change in systolic and diastolic blood pressure | Baseline to week 28
  Measured in millimeters of mercury (mmHg).
Number of Treatment Emergent Adverse Events (TEAEs) | Baseline to end of study (week 34)
  Count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com